CLINICAL TRIAL: NCT05947253
Title: Comparative Effects of BBT and Active Cycle of Breathing Technique on Dyspnea and Quality of Life in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0318
Record Dates: First submitted 2023-06-14; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: COPD
Keywords: Buteyko breathing technique
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: make 2 groups Patients who will meet the inclusion criteria will be recruited by convenient sampling technique and allocated in two groups by simple randomization process. First Group A 20 participants received Buyteko breathing technique while Group B 20 participants received active cycle of breathing technique and session of 35min will be given 5 days per week and data will be collected by using St. George's respiratory questionnaire for determining the quality of life and Borg's dyspnea scale for measuring breathlessness.
Who Masked: Participant, Investigator
Masking Description: Group A 20 participants received Buyteko breathing technique while Group B 20 participants received active cycle of breathing technique and session of 35min will be given 5 days per week and data will be collected by using St. George's respiratory questionnaire for determining the quality of life and Borg's dyspnea scale for measuring breathlessness. participant and investigator are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUTYEKO BREATHING TECHNIQUE (Experimental): First Group A 20 participants received Buyteko breathing technique while will be given 5 days per week
  Interventions: Other: Buyteko breathing technique
- active cycle of breathing technique (Experimental): Group B 20 participants received active cycle of breathing technique and session of 35min will be given 5 days per week
  Interventions: Other: active cycle of breathing technique

INTERVENTIONS:
Other: Buyteko breathing technique — group A 20 participants received Buyteko breathing technique 2 session for 3 weeks
  Arms: BUTYEKO BREATHING TECHNIQUE
Other: active cycle of breathing technique — Group B 20 participants received active cycle of breathing technique 2 session for 3 weeks
  Arms: active cycle of breathing technique

SUMMARY:
Comparative effects of Butyeko breathing technique and Active Cycle of Breathing technique on dyspnea and quality of life in patients with chronic obstructive pulmonary disease

DETAILED DESCRIPTION:
A comparative study to determine the effects of butyeko breathing techniques and Active Cycle of Breathing technique on dyspnea and quality of life in patients with chronic obstructive pulmonary disease. As few researches on Butyeko breathing techniques are still present on COPD most of them are on asthma. The goal of the Butyeko Method is to improve breathing patterns, as indicated by achieving a higher breath hold time (control pause). Every five seconds improvement to the control pause, results in an alleviation of breathing difficulty and improved control of COPD The Butyeko method is a purported method of "retraining" the body's breathing pattern to correct for the presumed chronic hyperventilation and hypocapnea, and thereby treat or cure the body of these medical problems. Patients with chronic obstructive pulmonary disease (COPD) often suffer from expectoration. To address this problem, active cycle of breathing techniques (ACBT) can be applied in patients of COPD. In our study daily Butyeko breathing exercise and active cycle of breathing technique session of 30 to 35 minutes will be given to patients and effects of both techniques will be compared.

A randomized clinical trial will be conducted using convenient sampling or randomized sampling technique in population of chronic obstructive pulmonary disease (COPD).Total sample size will be of 40 and two Groups will be made Group A 20 participants received Buyteko breathing technique and Groups B 20 participants received Active cycle of breathing technique. Data will be collected by using Borg's dyspnea scale, St.George Respiratory questionnaire and by pulmonary function testing. Data will be collected from pulmonary ward Jinnah hospital Lahore whole study will take total duration of 10 months and data will be analyzed using latest version of SPSS-25 software.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD confirmed by smoking history.
* PFT showing irreversible airflow limitation.
* Patients hemodynamically stable.
* Males and females.
* Patients capable of completing IPAQ questionnaire

Exclusion Criteria:

* Evidence of unstable cardiac disease, Pulmonale decompensation
* Disabling diseases which prevented participation in the exercise program, such as orthopedic inabilities or peripheral vascular disease.
* Systemic illness.
* Resting O2 saturation <90% with room air breathing and Patient with viral infection

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Borg's dyspnea scale. | 4 weeks
  For the measurement of dyspnea The Modified Borg Dyspnea Scale (MBS) is a 0 to 10 rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise and is routinely administered during six-minute walk testing (6MWT
Spirometry | 4 weeks
  Spirometry is the most common of the pulmonary function tests. It measures lung function, specifically the amount and/or speed of air that can be inhaled and exhaled.
  Spirometry is helpful in assessing breathing patterns that identify conditions such as asthma, Chronic obstructive pulmonary disease

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Principal Investigator — Riphah International University
Locations (1):
- Pulmonary ward Jinnah hospital Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogelmeier CF, Roman-Rodriguez M, Singh D, Han MK, Rodriguez-Roisin R, Ferguson GT. Goals of COPD treatment: Focus on symptoms and exacerbations. Respir Med. 2020 May;166:105938. doi: 10.1016/j.rmed.2020.105938. Epub 2020 Mar 21. PMID 32250871
- [Background] May SM, Li JT. Burden of chronic obstructive pulmonary disease: healthcare costs and beyond. Allergy Asthma Proc. 2015 Jan-Feb;36(1):4-10. doi: 10.2500/aap.2015.36.3812. PMID 25562549
- [Background] Halpin DM, Miravitlles M. Chronic obstructive pulmonary disease: the disease and its burden to society. Proc Am Thorac Soc. 2006 Sep;3(7):619-23. doi: 10.1513/pats.200603-093SS. PMID 16963544
- [Background] Fazleen A, Wilkinson T. Early COPD: current evidence for diagnosis and management. Ther Adv Respir Dis. 2020 Jan-Dec;14:1753466620942128. doi: 10.1177/1753466620942128. PMID 32664818
- [Background] Smith MC, Wrobel JP. Epidemiology and clinical impact of major comorbidities in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2014 Aug 27;9:871-88. doi: 10.2147/COPD.S49621. eCollection 2014. PMID 25210449
- [Background] Lopez AD, Shibuya K, Rao C, Mathers CD, Hansell AL, Held LS, Schmid V, Buist S. Chronic obstructive pulmonary disease: current burden and future projections. Eur Respir J. 2006 Feb;27(2):397-412. doi: 10.1183/09031936.06.00025805. No abstract available. PMID 16452599